CLINICAL TRIAL: NCT03919422
Title: Effectiveness of Additional Thoracic Paravertebral Block in Improving Anesthetic Effects of Regional Anesthesia for Proximal Humeral Fracture Surgery in Elderly Patients: Study Protocol for a Randomized Controlled Trial
Brief Title: Paravertebral Block for Proximal Humeral Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaofeng WANG, Principal Investigator, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-030
Record Dates: First submitted 2019-04-14; First posted 2019-04-18 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Proximal Humeral Fracture
Keywords: thoracic paravertebral block; regional anesthesia; elderly; proximal humeral fracture; brachial plexus block; cervical plexus block; intercostobrachial nerve
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IC group (Active Comparator): Interscalene brachial plexus-Cervical plexus
  Interventions: Procedure: interscalene brachial plexus block and superficial cervical plexus block
- ICTP group (Experimental): Interscalene brachial plexus-Cervical plexus combined with T2 Paravertebral blockade
  Interventions: Procedure: T2 paravertebral block; Procedure: interscalene brachial plexus block and superficial cervical plexus block

INTERVENTIONS:
Procedure: T2 paravertebral block — Ultrasound guided T2 thoracic paravertebral block is added in ICTP group. After interscalene brachial plexus block and superficial cervical plexus block have been administrated, selective 2nd thoracic nerve root(T2) will be blocked with 10 ml of 0.25% ropivacaine(naropin).
  Other Names: T2 PVB(paravertebral blockade )
  Arms: ICTP group
Procedure: interscalene brachial plexus block and superficial cervical plexus block — An ultrasound-guided IC block using an ultrasound machine (Sonosite, USA), and an linear array probe with a sterile cover and a 22G(Gauge) block needle is performed. An in-plane approach, advancing the needle along the longitudinal axis of the ultrasound transducer and visualizing the entire shaft is employed. Twenty ml of 0.375% ropivacaine(naropin) is injected around brachial plexus and 10 ml of 0.25% ropivacaine around superficial cervical plexus.
  Other Names: IC block

SUMMARY:
This study evaluates the effects of T2 paravertebral block block improving interscalene brachial plexus block and superficial cervical plexus block on the relief of pain intensity during elderly proximal humerus fracture fixation surgery. The brachial plexus and cervical plexus block(IC block) will be performed in half of participants, while the T2 paravertebral block combined with IC block will be performed in the other half.

ELIGIBILITY:
Inclusion Criteria:

1. Participant age≥ 65 years
2. Body mass index (BMI) < 30kg/m2
3. American Society of Anesthesiologists (ASA) classification I-II
4. Anterior operative incision approach

Exclusion Criteria:

1. Request for general anesthesia
2. Nerve block is unable to be performed due to various reasons
3. Coagulation dysfunction or anticoagulation therapy
4. History of upper limb nerve injury or phrenic nerve injury
5. Multiple trauma
6. Uncontrolled respiratory disease (severe chronic obstructive pulmonary disease, asthma, pulmonary infection, pneumothorax, etc.)
7. Uncontrolled hypertension (systolic pressure over 180mmHg or diastolic pressure over 110mmHg)
8. Uncontrolled heart disease (coronary heart disease, valvular disease or arrhythmia, etc.)
9. Stroke or cognitive dysfunction (unable to communicate or cooperate)
10. Hypersensitivity or allergy to anesthetics (ropivacaine or remifentanil)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang X, Zhang H, Chen Y, Zhang Q, Xie Z, Liao J, Jiang W, Zhang J. Is It Useful and Necessary to Add a T2 Paravertebral Block to the Regional Anesthesia During Proximal Humeral Fracture Surgery in Elderly Patients? A Prospective and Randomized Controlled Trial. Front Surg. 2022 Mar 14;9:755298. doi: 10.3389/fsurg.2022.755298. eCollection 2022. PMID 35360431
- [Derived] Wang X, Zhang H, Xie Z, Zhang Q, Jiang W, Zhang J. The effectiveness of additional thoracic paravertebral block in improving the anesthetic effects of regional anesthesia for proximal humeral fracture surgery in elderly patients: study protocol for a randomized controlled trial. Trials. 2020 Feb 19;21(1):204. doi: 10.1186/s13063-020-4078-9. PMID 32075674

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 121participants were screened. 41 did not meet criteria.
Period: Overall Study
Arm/Group | IC Group | ICTP Group
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IC Group | ICTP Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (6.0) | 74.5 (6.5) | 74.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 62
  Male | 6 | 12 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  yellow race, Han nationality, China | 40 | 40 | 80
weight [Mean (Standard Deviation); unit: kg] | 60.2 (9.1) | 62.5 (11.3) | 61.3 (10.3)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (3.2) | 24.4 (3.8) | 24.4 (3.5)
ASA [Count of Participants; unit: Participants] — The ASA risk classification system can be used to quantify the risk associated with anesthesia and surgery. ASA I: Healthy patient without organic, biochemical, or psychiatric disease. ASA II: A patient with mild systemic disease. ASA III: Significant or severe systemic disease that limits normal activity. ASA IV: Severe disease that is a constant threat to life or requires intensive therapy. ASA V: Moribund patient who is equally likely to die in the next 24 hours with or without surgery. ASA VI: Brain-dead organ donor.
  Participants
    ASA I | 14 | 17 | 31
    ASA II | 26 | 23 | 49
duration of surgery [Median (Inter-Quartile Range); unit: minutes] | 72.5 [46.3 to 93.8] | 70 [56.3 to 90] | 70 [51.3 to 90]
height [Mean (Standard Deviation); unit: cm] | 157.2 (6.8) | 159.7 (7.2) | 159.7 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Success Rate(Ability to Proceed With Surgery Without the Need for Intravenous Narcotics, General Anaesthesia, Rescue Blocks or Local Infiltration by the Surgeon)
Description: Success rate - was equivalent to surgical anesthesia, defined as the ability to proceed with surgery without the need for intravenous narcotics, general anaesthesia, rescue blocks or local infiltration by the surgeon.
Time Frame: throughout the operation duration, an average of 2 to 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IC Group | ICTP Group
Number analyzed (Participants) | 40 | 40
Participants | 31 | 21

2. Secondary Outcome: Assessment of Sensory Blockade
Description: Sensory blockade graded from 0 to 2(0= normal sensation, 1= decreased sensation and 2= no perception) by applying pinprick and cold test to the different parts of shoulder
Time Frame: 20 minutes after all the nerve block operations have been finished
Measure: Count of Participants; unit: Participants
Arm/Group | IC Group | ICTP Group
Number analyzed (Participants) | 40 | 40
Participants
  distal clavicle area: no block | 1 | 0
  distal clavicle area: partial block | 2 | 1
  distal clavicle area: complete block | 37 | 39
  deltoid area: no block | 0 | 0
  deltoid area: partial block | 3 | 2
  deltoid area: complete block | 37 | 38
  lateral part of upper arm: no block | 0 | 0
  lateral part of upper arm: partial block | 4 | 3
  lateral part of upper arm: complete block | 36 | 37
  medial part of upper arm: no block | 36 | 6
  medial part of upper arm: partial block | 4 | 17
  medial part of upper arm: complete block | 0 | 17

3. Secondary Outcome: Proportion of Participants Completed the Procedure With Remifentanil
Description: When the primary outcome of the participant is assessed by "failure" during the surgery, 0.25μg/kg/min remifentanil will be given via intravenous infusion. Two minutes later, the procedure will continue if the participant can tolerate the pain.
Time Frame: throughout the operation duration, an average of 2 to 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IC Group | ICTP Group
Number analyzed (Participants) | 40 | 40
Participants | 13 | 7

4. Secondary Outcome: Proportion of Participants Conversed Into General Anesthesia(Laryngeal Mask Airway,LMA)
Description: When the primary outcome of the participant is assessed by "failure" during the surgery, 0.25μg/kg/min remifentanil will be given via intravenous infusion. Two minutes later, if the participant cannot tolerate the pain, a general anesthesia with LMA will be given.
Time Frame: throughout the operation duration, an average of 2 to 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IC Group | ICTP Group
Number analyzed (Participants) | 40 | 40
Participants | 6 | 2

5. Secondary Outcome: Cumulative Doses of Intraoperative Vasoactive Medications (Urapidil,Atropine, Ephedrine)
Description: Cumulative doses of vasoactive drugs required such as urapidil,atropine, ephedrine during the surgery.
Time Frame: At the end of surgical procedure(an average of 2 to 3 hours)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | IC Group | ICTP Group
Number analyzed (Participants) | 40 | 40
mg
  urapidil (mg) | 1.13 (2.9) | 1.50 (3.6)
  atropine (mg) | 0.05 (0.2) | 0.09 (0.2)
  ephedrine (mg) | 1.00 (3.3) | 0.5 (2.2)

6. Secondary Outcome: Cumulative Doses of Intraoperative Vasoactive Medications (Deoxyepinephrine)
Description: Cumulative doses of intravenous deoxyepinephrine required during the surgery.
Time Frame: At the end of surgical procedure(an average of 2 to 3 hours)
Measure: Mean (Standard Deviation); unit: ug
Arm/Group | IC Group | ICTP Group
Number analyzed (Participants) | 40 | 40
ug | 5.0 (18.9) | 7.5 (29.0)

7. Secondary Outcome: Complications Related With Anesthesia
Description: Presence or absence of local anesthetic systemic toxicity, pneumothorax, and epidural block, total spinal block, hematoma
Time Frame: within 24 hours since the nerve block finished
Measure: Count of Participants; unit: Participants
Arm/Group | IC Group | ICTP Group
Number analyzed (Participants) | 40 | 40
Participants
  local anesthetic systemic toxicity | 0 | 0
  pneumothorax | 0 | 0
  epidural block | 0 | 0
  total spinal block | 0 | 0
  hematoma | 0 | 0

8. Secondary Outcome: Intraoperative Adverse Reactions (Including Hypertension, Hypotension, Bradycardia, Tachycardia or Dyspnea)
Description: Number of participants with hypertension, hypotension, bradycardia, tachycardia or dyspnea during the surgery.
Time Frame: throughout the operation duration, an average of 2 to 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | IC Group | ICTP Group
Number analyzed (Participants) | 40 | 40
Participants
  Number of participants with hypertension during the surgery | 6 | 7
  Number of participants with hypotension during the surgery | 4 | 5
  Number of participants with bradycardia during the surgery | 5 | 8
  Number of participants with tachycardia druing the surgery | 0 | 1
  Number of participants with dyspnea during the surgery | 5 | 2

ADVERSE EVENTS:
Time Frame: 1day after surgery
Description: Block-related complications such as local anesthetic systemic toxicity, pneumothorax, epidural block, total spinal block and hematoma were defined as Severe Adverse Events. The intraoperative adverse reactions including hypertension, hypotension, bradycardia, tachycardia and dyspnea were defined as Other Adverse Events.
Arm/Group | IC Group | ICTP Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 20/40 | 23/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC Group (N=40) | ICTP Group (N=40)
local anesthetic systemic toxicity (Nervous system disorders) | 0 (0) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
epidural block (Nervous system disorders) | 0 (0) | 0 (0)
total spinal block (Nervous system disorders) | 0 (0) | 0 (0)
hematoma (Vascular disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC Group (N=40) | ICTP Group (N=40)
Hypertension (Cardiac disorders) | 6 (6) | 7 (7)
hypotension (Cardiac disorders) | 4 (4) | 5 (5)
bradycardia (Cardiac disorders) | 5 (5) | 8 (8)
tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT03919422/Prot_SAP_000.pdf